CLINICAL TRIAL: NCT00773955
Title: A Phase II Study of AT-101 in Recurrent Extensive Stage Small Cell Lung Cancer
Brief Title: R-(-)-Gossypol Acetic Acid in Treating Patients With Recurrent Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01058; NCI-2009-01058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0721; CDR0000616965; MC0721 (Other: Mayo Clinic); 8027 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH); N01CM62209 (NIH); NCT01647113 (obsolete NCT alias)
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2011-10

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — gossypol acetic acid

ARMS (1):
- Treatment (R-(-)-gossypol) (Experimental): Patients receive oral R-(-)-gossypol once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: R-(-)-gossypol acetic acid; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: R-(-)-gossypol acetic acid — Given orally
  Other Names: AT-101
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well R-(-)-gossypol acetic acid works in treating patients with recurrent extensive-stage small cell lung cancer. Drugs used in chemotherapy, such as R-(-)-gossypol acetic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate of R-(-)-gossypol in patients with recurrent chemotherapy-sensitive extensive stage small cell lung cancer.

II. To determine the time to disease progression. III. To determine the overall survival. IV. To assess the toxicities associated with this drug. V. To explore whether intratumoral Bcl-2 family member expression correlates with sensitivity to targeting by R-(-)-gossypol.

VI. To explore whether the administration of R-(-)-gossypol causes specific induction of the intrinsic apoptotic pathway.

OUTLINE: This is a multicenter study.

Patients receive oral R-(-)-gossypol once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood is collected periodically during treatment for pharmacodynamic analysis. Peripheral blood mononuclear cells are analyzed via protein isolation and western blotting for Bcl-2, cytoplasmic release of cytochrome c, and caspase activation. Available tumor tissue blocks are assessed by immunohistochemistry.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer

  * Extensive stage disease
  * Recurrent disease
* Measurable disease
* Chemotherapy-sensitive disease, defined as:

  * No progression during first-line chemotherapy
  * No disease recurrence < 2 months after completion of first-line chemotherapy
* Must have received prior platinum-based chemotherapy
* No symptomatic or progressive brain metastases

  * Patients with previously treated brain metastases who are clinically and radiographically stable or improved and have been off steroids ≥ 14 days are eligible
* ECOG performance status 0-2
* Life expectancy > 12 weeks
* Leukocytes ≥ 3,000/μL
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin < 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Hemoglobin > 8 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 30 days after completion of study therapy
* Able to take oral medications on a regular basis
* Willing to provide blood samples for mandatory correlative studies
* No condition that impairs the ability to swallow and retain R-(-)-gossypol tablets, including the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Active peptic ulcer disease
* No malabsorption syndrome or disease significantly affecting gastrointestinal function
* No ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No symptomatic hypercalcemia > grade 2
* No requirement for routine use of hematopoietic growth factors (including G-CSF, GM-CSF, or IL-11) or platelet transfusions to maintain ANC or platelet counts
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to R-(-)-gossypol
* No HIV positivity
* Recovered from all prior therapy, including prior surgical procedures
* No prior surgical procedures affecting absorption
* No prior resection of the stomach or small bowel
* No more than one prior chemotherapy regimen
* No prior racemic gossypol or R-(-)-gossypol
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 4 weeks since prior radiotherapy, hormonal agents, or biologic response modifiers
* At least 4 weeks since prior and no concurrent investigational agents or devices
* No concurrent prophylactic hematopoietic growth factors (including filgrastim [G-CSF], sargramostim [GM-CSF], or interleukin-11 [IL-11]) during course one
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Baggstrom, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2008 to January 2010, 15 patients were accrued to the study from five sites within the Mayo Clinic Phase 2 Consortium and the California Consortium.
Pre-assignment Details: One patient discontinued therapy after one cycle of treatment due to persistent grade 1 thrombocytopenia. Therefore, fourteen patients were evaluable for the primary end point at the interim analysis. All 15 patients were included in secondary endpoint analysis.
Period: Overall Study
Arm/Group | Treatment (R-(-)-Gossypol)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (R-(-)-Gossypol)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 67.0 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14
  Australia | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Tumor Response Defined to be Either a Complete Response (CR) or Partial Response (PR)
Description: The number of successes will be estimated by counting the number of participants with confirmed responses. A confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions:
  A Complete Response (CR) requires the disappearance of all target lesions
  A Partial Response (PR) requires a >=30% decrease in the sum of the longest diameter of target lesions from baseline measurements.
Time Frame: During the first 6 courses of treatment
Population: One patient discontinued therapy after one cycle of treatment due to persistent grade 1 thrombocytopenia. Therefore, fourteen patients were evaluable for the primary end point at the interim analysis.
Measure: Number; unit: participants
Arm/Group | Treatment (R-(-)-Gossypol)
Number analyzed (Participants) | 14
participants
  Confirmed Partial Response (PR) | 0
  Confirmed Complete Response (CR) | 0

2. Secondary Outcome: Survival Time
Description: Estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 5 years
Population: All 15 patients were analyzed for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (R-(-)-Gossypol)
Number analyzed (Participants) | 15
months | 8.5 [8.1 to 10.2]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date documentation of disease progression. Estimated using the method of Kaplan-Meier.
  Per the RECIST criteria, progression is defined as at least a 20% increase in the sum of Longest Dimension (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From registration to the earliest date documentation of disease progression, assessed up to 5 years
Population: All 15 patients were analyzed for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (R-(-)-Gossypol)
Number analyzed (Participants) | 15
months | 1.7 [1.5 to 2.0]

4. Secondary Outcome: Duration of Response
Time Frame: From the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented, assessed up to 5 years
Population: There were no confirmed responses qualifying for this endpoint.
Arm/Group | Treatment (R-(-)-Gossypol)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (R-(-)-Gossypol)
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R-(-)-Gossypol) (N=15)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R-(-)-Gossypol) (N=15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (20)
Sinus tachycardia (Cardiac disorders) | 2 (7)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (13)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (6)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (17)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 3 (5)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 5 (7)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 5 (7)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 9 (12)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (7)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less